CLINICAL TRIAL: NCT00882297
Title: Subclavian Vein Ultrasound Guided Cannulation in Adult: Transversal and Longitudinal Approach Comparison
Brief Title: Subclavian Vein Ultrasound Guided Cannulation in Adult
Acronym: CATETEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHUBX 2009/06
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Cardiac Surgery
Keywords: Ultrasoundography; catheterization; central venous subclavian vein methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Transversal approach guided placement
  Interventions: Procedure: Echoguided vein puncture
- 2 (Active Comparator): Longitudinal approach guided placement
  Interventions: Procedure: Echoguided vein puncture

INTERVENTIONS:
Procedure: Echoguided vein puncture — Puncture with echographic visualization of vein in transversal and longitudinal way.

SUMMARY:
There is actually two techniques of subclavian vein ultrasonography-guided venous catheterization : the axial and longitudinal approach. Currently, nothing makes it possible to privilege one technique compared to the other. This study aims to determine the best ultrasonography-guided method.

DETAILED DESCRIPTION:
This prospective randomized study will concern 100 adult patients operated of cardiac surgery under general anesthesia and requiring a central venous catheter. Patients will be randomized by an operator experienced in echoguided venous catheterization to be included in the axial (50 patients) or the longitudinal (50 patients) approach group. The device used will be a vascular probe of 7.5 MHz (Sonosite I Look®). The principal outcome measure will be the time from percutaneous puncture to the rise of the metallic guide (seldinger technique). The secondary criteria will be the rate of complication and failure. A series of echographic (size and depth of the subclavian vein and biometric (BMI, theoretical distance not from puncture (way of Aubaniac)/réel) measurements will be done to identify predictive conditions of success or failure depending of the echographic approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring the installation of a central venous catheter in subclavian site
* Installation of catheter under general anaesthesia
* Oral consent of the patient

Exclusion Criteria:

* Thrombosis in subclavian vein
* Urgency of central venous catheterization.
* Insertion of central vein catheter other than subclavian
* Insertion of subclavian catheter under loco-regional anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Time from vein puncture to seldinger guide placement | After anesthesia during cardiac surgery

SECONDARY OUTCOMES:
Complications | During cardiac surgery until 48 hours after the end

CONTACTS AND LOCATIONS:
Overall Officials: Joachim CALDERON, MD, Principal Investigator — University Hospital, Bordeeaux
Locations (1):
- University Hospital, Bordeaux, Pessac, France

REFERENCES:
- [Background] Taylor RW, Palagiri AV. Central venous catheterization. Crit Care Med. 2007 May;35(5):1390-6. doi: 10.1097/01.CCM.0000260241.80346.1B. PMID 17414086
- [Background] Forestier F, Rossi H, Calderon J, Soubiron L, Bourdarias B, Janvier G. [Training for adult subclavian venous catheterization: use of real-time echography]. Ann Fr Anesth Reanim. 2002 Nov;21(9):698-702. doi: 10.1016/s0750-7658(02)00778-5. French. PMID 12494802
- [Background] Brooks AJ, Alfredson M, Pettigrew B, Morris DL. Ultrasound-guided insertion of subclavian venous access ports. Ann R Coll Surg Engl. 2005 Jan;87(1):25-7. doi: 10.1308/1478708051441. PMID 15720903